CLINICAL TRIAL: NCT01892995
Title: Ketamine for Acute Suicidal Ideation in the Emergency Department: Randomized Controlled Trial
Acronym: LDK-SI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Brooke Army Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Steven Schauer, CPT, Brooke Army Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BAMC-385833-1; NCT02367586 (obsolete NCT alias)
Record Dates: First submitted 2013-07-02; First posted 2013-07-08 (Estimated); Last update posted 2015-02-16 (Estimated); Status verified 2015-02

CONDITIONS: Suicide
Keywords: suicide; ketamine; low-dose ketamine; suicidal ideations; emergency department
MeSH Terms: conditions — Suicide; Suicidal Ideation; Emergencies | interventions — Ketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Ketamine (Experimental): active arm
  Interventions: Drug: Ketamine
- Diphenhydramine (Sham Comparator): sham arm
  Interventions: Drug: Ketamine
- Saline (Placebo Comparator): placebo
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Ketamine

SUMMARY:
This study will enroll patients presenting to the emergency department with acute suicidal ideation meeting inclusion and exclusion criteria. Patients will be randomized to one of three arms: ketamine (intervention) or diphenhydramine (control) or placebo (control). Serial measurements will be made in the ED and at follow-up intervals.

ELIGIBILITY:
Inclusion Criteria:

* Patients age 18 to less than 75 who present to the SAMMC ED with either overt or incidental suicidal ideations with a SADPERSONS score 5 or greater that the treating provider feels warrant formal evaluation.

Exclusion Criteria:

* -Poor vital sign stability hypoxia: O2 < 95%, hypotension: SBP< 90 hypertension: SBP>180 Heart rate: < 50 or >120 Respiratory Rate: <10 or >30
* Altered mental status or intoxication
* Patient is unwilling to participate or provide informed consent
* Any allergy to ketamine or diphenhydramine
* Patient is female of child-bearing age and unwilling to provide urine or blood for HCG analysis
* Pregnancy or breast feeding
* Presence of chronic oxygen-dependent pulmonary disease, liver cirrhosis, or renal disease requiring dialysis
* Presence of ischemic heart disease, heart failure, or a history of unstable dysrhythmias
* Presence of intracranial mass or vascular lesion.
* Presence of a history of psychosis or hallucinations (as assessed by electronic chart review)
* Weight greater than 115 kg or less than 45kg
* History of increased intracranial pressure/hypertensive hydrocephalus
* Non-English speaking patients
* Patient is acutely psychotic
* Provider feels that patient currently or likely will require chemical and/or physical restraints
* History of prolonged QT-interval

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 53 (Estimated)
Dates: Start 2015-06; Primary Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Change in Beck Scale for Suicidal Ideation | 2 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Brooke Army Medical Center, Fort Sam Houston, Texas, United States